CLINICAL TRIAL: NCT02462434
Title: Impact of Early Intervention on Maternal Stress in Mothers of Fetuses Diagnosed With Single Ventricle Physiology Requiring Neonatal Surgery
Brief Title: Impact of Early Intervention on Maternal Stress in Mothers of Fetuses Diagnosed With Single Ventricle Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Karen Uzark, Associate Professor of Cardiac Surgery and Associate Professor of Pediatric Cardiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00072957
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Single Ventricle Defect; Stress, Psychological
Keywords: Pediatric palliative care
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Univentricular Heart; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early palliative care team consultation (Experimental): Early pediatric palliative care team consultation for single ventricle patients will occur in this group following birth but prior to the first stage palliative surgery.
  Interventions: Behavioral: Early palliative care team consultation
- Usual care (No Intervention): Usual care for single ventricle patients will be provided with palliative care team consultation occurring at any point (if it is determined the child and family would benefit from palliative care consultation) during the child's neonatal hospital stay.

INTERVENTIONS:
Behavioral: Early palliative care team consultation — The palliative care team will evaluate the patient and family with the following core palliative care goals in mind: evaluating maternal understanding of their child's diagnosis and eliciting maternal concerns regarding their child's physical symptoms, identifying maternal social support systems and additional life stressors, identifying maternal expectations and hopes for their child's medical care, and assessing maternal fears surrounding their child's diagnosis and medical treatments. Palliative care team support and resources will then be provided in areas of necessity identified for the family. Palliative care team follow up will then be determined based on the level of need identified for each individual study participant.
  Arms: Early palliative care team consultation

SUMMARY:
This study evaluates maternal psychological distress and the impact of early palliative care team consultation on maternal anxiety and depression symptoms, coping, and quality of life/family functioning in the care of neonates born with single ventricle physiology. Half of the participants will receive early palliative care team consultation, while the other half will receive usual care (no or late palliative care intervention). The investigators hypothesize maternal stress, anxiety, and depression will be lower in the palliative care intervention group compared with the control group, and maternal coping mechanisms and perceived quality of life and family functioning will improve at the pre-discharge assessment.

DETAILED DESCRIPTION:
Mothers of children with congenital heart disease are at increased risk of psychological morbidity including stress, anxiety, and depression. In particular, mothers of patients with single ventricle physiology who require neonatal surgery, face a great deal of stress related to the risk of serious complications including neonatal death. Previous studies have suggested that providing emotional psychosocial support may modify the development of significant psychosocial problems in parents of children with congenital heart disease. The pediatric palliative care team specializes in multiple elements of psychological and spiritual care for families of such children.

The purpose of this pilot study is to evaluate maternal psychological distress and to examine the potential impact of early palliative care team consultation on maternal anxiety and depression symptoms, coping, and quality of life/family functioning in the care of neonates born with single ventricle physiology. Mothers will complete four questionnaires measuring anxiety, depression, and quality of life/family functioning at a prenatal follow up visit and again prior to neonatal surgical hospital stay discharge (or at 30 days). Infants will be randomly assigned (by date of birth) to receive early palliative care team consultation or usual care (no or late palliative care intervention).

The investigators hypothesize maternal stress, anxiety, and depression will be lower in the palliative care intervention group compared with the control group, and maternal coping mechanisms and perceived quality of life and family functioning will improve at the pre-discharge assessment.

ELIGIBILITY:
Inclusion Criteria:

* Mothers pregnant with fetuses with single ventricle physiology who are planned to undergo staged single ventricle palliative surgery with the first surgery occurring in the neonatal period.

Exclusion Criteria:

* Mothers with neonates born at a gestational age of less than 32 weeks requiring admission and management in the Neonatal Intensive Care Unit.
* Mothers with neonates diagnosed with major non-cardiac congenital anomalies requiring additional surgical management beyond cardiac surgery in the neonatal period.
* Non-English-speaking mothers who are unable to adequately comprehend and respond to survey questions administered as part of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10-12 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Change in maternal State-Trait Anxiety Index scores | Up to 4 weeks
  Mothers will complete the State-Trait Anxiety Index to assess current anxiety symptoms and trait-like anxiety symptoms (with clinical cut-off scores defined when applicable) at a prenatal follow up visit and again prior to neonatal surgery discharge.
Change in maternal Beck Depression Index II scores | Up to 4 weeks
  Mothers will complete the Beck Depression Index II to assess severity of depressive symptoms (with clinical cut-off scores defined when applicable) at a prenatal follow up visit and again prior to neonatal surgery discharge.
Change in maternal Brief Cope Inventory survey scores | Up to 4 weeks
  Mothers will complete the Brief Cope Inventory to assess a broad range of coping responses (with clinical cut-off scores defined when applicable) at a prenatal follow up visit and again prior to neonatal surgery discharge.
Change in maternal PedsQL Family Impact Module survey scores | Up to 4 weeks
  Mothers will complete the PedsQL Family Impact Module to measure the impact of the child's cardiac diagnosis on the parents and family to indicate parent functioning and overall family functioning (with clinical cut-off scores defined when applicable) at a prenatal follow up visit and again prior to neonatal surgery discharge.

SECONDARY OUTCOMES:
Length of neonate's intensive care unit (ICU) stay in days | Participants will be followed for the duration of ICU stay, an expected average of 2 weeks
  Continuous days of initial ICU stay from time of admission
Length of neonate's total hospital stay in days | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Continuous acute care inpatient hospital days from day of admission until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hayley S Hancock, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Lawoko S, Soares JJ. Psychosocial morbidity among parents of children with congenital heart disease: a prospective longitudinal study. Heart Lung. 2006 Sep-Oct;35(5):301-14. doi: 10.1016/j.hrtlng.2006.01.004. PMID 16963362
- [Background] Rychik J, Donaghue DD, Levy S, Fajardo C, Combs J, Zhang X, Szwast A, Diamond GS. Maternal psychological stress after prenatal diagnosis of congenital heart disease. J Pediatr. 2013 Feb;162(2):302-7.e1. doi: 10.1016/j.jpeds.2012.07.023. Epub 2012 Sep 10. PMID 22974576
- [Background] Uzark K, Jones K. Parenting stress and children with heart disease. J Pediatr Health Care. 2003 Jul-Aug;17(4):163-8. doi: 10.1067/mph.2003.22. PMID 12847425
- [Background] Helfricht S, Latal B, Fischer JE, Tomaske M, Landolt MA. Surgery-related posttraumatic stress disorder in parents of children undergoing cardiopulmonary bypass surgery: a prospective cohort study. Pediatr Crit Care Med. 2008 Mar;9(2):217-23. doi: 10.1097/PCC.0b013e318166eec3. PMID 18477936
- [Background] Sarajuuri A, Lonnqvist T, Schmitt F, Almqvist F, Jokinen E. Patients with univentricular heart in early childhood: parenting stress and child behaviour. Acta Paediatr. 2012 Mar;101(3):252-7. doi: 10.1111/j.1651-2227.2011.02509.x. Epub 2011 Nov 29. PMID 22040350
- [Background] Vrijmoet-Wiersma CM, Ottenkamp J, van Roozendaal M, Grootenhuis MA, Koopman HM. A multicentric study of disease-related stress, and perceived vulnerability, in parents of children with congenital cardiac disease. Cardiol Young. 2009 Dec;19(6):608-14. doi: 10.1017/S1047951109991831. Epub 2009 Oct 14. PMID 19825253
- [Background] Ohye RG, Schonbeck JV, Eghtesady P, Laussen PC, Pizarro C, Shrader P, Frank DU, Graham EM, Hill KD, Jacobs JP, Kanter KR, Kirsh JA, Lambert LM, Lewis AB, Ravishankar C, Tweddell JS, Williams IA, Pearson GD; Pediatric Heart Network Investigators. Cause, timing, and location of death in the Single Ventricle Reconstruction trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):907-14. doi: 10.1016/j.jtcvs.2012.04.028. Epub 2012 Aug 15. PMID 22901498
- [Background] Ohye RG, Sleeper LA, Mahony L, Newburger JW, Pearson GD, Lu M, Goldberg CS, Tabbutt S, Frommelt PC, Ghanayem NS, Laussen PC, Rhodes JF, Lewis AB, Mital S, Ravishankar C, Williams IA, Dunbar-Masterson C, Atz AM, Colan S, Minich LL, Pizarro C, Kanter KR, Jaggers J, Jacobs JP, Krawczeski CD, Pike N, McCrindle BW, Virzi L, Gaynor JW; Pediatric Heart Network Investigators. Comparison of shunt types in the Norwood procedure for single-ventricle lesions. N Engl J Med. 2010 May 27;362(21):1980-92. doi: 10.1056/NEJMoa0912461. PMID 20505177
- [Background] Morell E, Wolfe J, Scheurer M, Thiagarajan R, Morin C, Beke DM, Smoot L, Cheng H, Gauvreau K, Blume ED. Patterns of care at end of life in children with advanced heart disease. Arch Pediatr Adolesc Med. 2012 Aug;166(8):745-8. doi: 10.1001/archpediatrics.2011.1829. PMID 22473887
- [Background] Himelstein BP, Hilden JM, Boldt AM, Weissman D. Pediatric palliative care. N Engl J Med. 2004 Apr 22;350(17):1752-62. doi: 10.1056/NEJMra030334. No abstract available. PMID 15103002
- [Background] Mack JW, Wolfe J. Early integration of pediatric palliative care: for some children, palliative care starts at diagnosis. Curr Opin Pediatr. 2006 Feb;18(1):10-4. doi: 10.1097/01.mop.0000193266.86129.47. PMID 16470155
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Ayers S. Assessing psychopathology in pregnancy and postpartum. J Psychosom Obstet Gynaecol. 2001 Jun;22(2):91-102. doi: 10.3109/01674820109049959. PMID 11446159
- [Background] Medrano GR, Berlin KS, Hobart Davies W. Utility of the PedsQL family impact module: assessing the psychometric properties in a community sample. Qual Life Res. 2013 Dec;22(10):2899-907. doi: 10.1007/s11136-013-0422-9. Epub 2013 Apr 27. PMID 23625591